CLINICAL TRIAL: NCT06742437
Title: Efficacy and Safety of a New Sperm Capacitation Method: a Prospective in Vitro Study on Semen Samples
Brief Title: Efficacy and Safety of a New Sperm Capacitation Method
Acronym: HyperSperm01
Status: Recruiting | Type: Observational
Sponsor: Fecundis Lab SL (Other)
Responsible Party: Sponsor
Other Study IDs: HyperSperm01
Record Dates: First submitted 2024-12-12; First posted 2024-12-19 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Reproductive Issues; Male Infertility; Asthenozoospermia; Oligozoospermia; Teratozoospermia
MeSH Terms: conditions — Infertility, Male; Asthenozoospermia; Oligospermia; Teratozoospermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Normozoospermic: Semen samples with normal sperm parameters as defined by the World Health Organization guidelines (e.g., normal sperm concentration, motility, and morphology).
  Interventions: Device: Standard sperm preparation; Device: HyperSperm
- Teratozoospermic: Semen samples with abnormal sperm morphology, where the percentage of morphologically normal sperm is below the threshold set by the World Health Organization (i.e., 4%).
  Interventions: Device: Standard sperm preparation; Device: HyperSperm
- Asthenozoospermic: Semen samples characterized by reduced sperm motility, where the percentage of progressive motile sperm is below the threshold set by the World Health Organization (i.e., 32%).
  Interventions: Device: Standard sperm preparation; Device: HyperSperm
- Oligozoospermic: Semen samples with a low sperm concentration, below the World Health Organization reference value (i.e., less than 15 million sperm per milliliter).
  Interventions: Device: Standard sperm preparation; Device: HyperSperm
- Cryopreserved semen: Semen samples that have been preserved through freezing and stored at ultra-low temperatures.
  Interventions: Device: Standard sperm preparation; Device: HyperSperm

INTERVENTIONS:
Device: Standard sperm preparation — Sperm samples in the control group will undergo traditional processing
Device: HyperSperm — Sperm samples in the experimental group will undergo product-specific processing

SUMMARY:
Prospective, multicenter research study with a split-sample design on semen samples, without intervention, to evaluate the efficacy and safety of HyperSperm, a new sperm capacitation method, in 300 semen samples with various characteristics and abnormalities, in an in vitro study over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide a semen sample via masturbation

Exclusion Criteria:

* Current diagnosis of a sexually transmitted infection (STI)
* Previous diagnosis of hepatitis A, B, C, D, or HIV
* Prior participation in this study
* Participation in a clinical trial involving an intervention within the last 3 months

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Men attending fertility clinics who provide a semen sample with normal parameters (normozoospermia), or present a male factor (asthenozoospermia, oligozoospermia, teratozoospermia, or a combination thereof).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Hyperactivation | 2 hours
  Percentage of sperm cells displaying hyperactivated motility

SECONDARY OUTCOMES:
Sperm vitality | 2 hours
  Percentage of viable sperm cells
DNA fragmentation | 2 hours
  Percentage of TUNEL-positive sperm cells
Sperm motility | 2 hours
  Percentage of motile sperm cells
Survival | 20 hours
  Percentage of motile sperm cells after overnight incubation

CONTACTS AND LOCATIONS:
Overall Officials: Mariona Rius Mas, PhD, Principal Investigator — Fertty
Locations (4):
- Spain (4):
  - Eugin Barcelona, Barcelona, Barcelona
  - Fertty, Barcelona, Barcelona
  - CIRH, Barcelona, Barcelona
  - Natuvitro, Barcelona, Barcelona